CLINICAL TRIAL: NCT03643757
Title: Comparison of Thoracic Epidural and Intravenous Analgesia From the Perspective of Recovery of Respiratory Function at Early Post-thoracotomy Period in Lung Cancer Surgery
Brief Title: Epidural Analgesia and Postoperative Respiratory Functions (EPAPRES)
Acronym: EPAPRES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yedikule Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Derya Ozden Omaygenc, Principal investigator, Yedikule Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2866
Record Dates: First submitted 2018-08-16; First posted 2018-08-23 (Actual); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Respiration Disorders
Keywords: Blood gas analysis; Epidural analgesia; Lung cancer; Respiratory function tests; Thoracotomy
MeSH Terms: conditions — Respiration Disorders; Lung Neoplasms | interventions — Tea; Bupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thoracic Epidural Analgesia (Active Comparator): Population to whom thoracic epidural analgesia with bupivacaine as a component of multimodal analgesia was administered.
  Interventions: Procedure: Thoracic epidural analgesia; Drug: Bupivacaine
- Intravenous analgesia (Active Comparator): Population to whom combined intravenous analgesia was administered.
  Interventions: Procedure: Thoracic epidural analgesia

INTERVENTIONS:
Procedure: Thoracic epidural analgesia — Before the initiation of the procedure, in the intervention group epidural catheter was inserted by loss of resistance method at the level of T3-T7 with the help of an 18 G Thuohy needle (Pajunk, Geisingen, Germany) while the patient was on sitting position. A test dose of 2 ml, 2% Lidocaine HCL was administered through the catheter. Once, efficacy was confirmed, 10 ml bolus dose of 0.1% Bupivacaine was injected. Analgesia maintenance was provided by infusion of 0.1% Bupivacaine (0.1 ml/kg/hour) both intra- and postoperatively for 24 hours.
  Other Names: Posterolateral thorachotomy; Intercostal blockade
Drug: Bupivacaine — In addition to multimodal analgesia protocol, epidural bupivacaine was administered in TEA arm and pain relief was achieved by intravenous pethidine infusion in IVA arm.
  Other Names: Pethidine intravenous infusion
  Arms: Thoracic Epidural Analgesia

SUMMARY:
Patients operated with posterolateral thoracotomy were enrolled. Post-operative analgesia was provided either by TEA with 0.1% bupivacaine or pethidine based intravenous analgesia (IVA) in our sample population. Perception of pain was quantified by Visual Analogue Scale (VAS) at rest and during coughing. Arterial blood samples were collected at 1st, 24th and 72nd hours of post-operative period. Pre-operative and post-operative 72nd-hour spirometric measurements were recorded

DETAILED DESCRIPTION:
lung cancer patients (between ages 18 to 75 and American Society of Anesthesiologists -ASA- Class I to III), undergoing an elective thoracic surgical procedure with posterolateral thoracotomy, were enrolled. The study was approved by the local ethical committee in Yedikule Chest Diseases and Thoracic Surgery Ed. and Research Hospital and therefore had been performed in accordance with global ethical standards. Written informed consent was received from all participants.

Individuals beyond defined age limits, patients who have psychiatric problems, auditory deficit, drug abuse, severe cardiovascular system disorders or severe respiratory depression depicted as having less than 50% of the predicted value of forced expiratory volume were excluded. Patients refusing to give consent and to whom inserting an epidural catheter is contraindicated were not involved either. Surgical procedures were performed by the same team. In the operating room, if serratus anterior muscle could not be spared or chest wall resection was performed, these patients were also excluded even though they had met other qualifications. Finally, patients who could not be extubated before transfer were not involved.

Regarding pre-operative evaluation, age, gender, weight, height, smoking status (package/years) and ASA score of patients were recorded.

For assessing the impact of method of analgesia on target parameters, patients were allocated to TEA and intravenous analgesia (IVA) groups. Randomisation was performed by closed envelope method.

2.2 Features of anesthetic technique and intraoperative analgesia Before the initiation of procedure, in TEA group epidural catheter was inserted by loss of resistance method at the level of T3-T7 with the help of a 18 G Thuohy needle (Pajunk, Geisingen, Germany) while patient was on sitting position. A test dose of 2 ml, 2% Lidocaine HCL was administered through the catheter. Once, efficacy was confirmed, 10 ml bolus dose of 0.1% Bupivacaine was injected. Analgesia maintanence was provided by infusion of 0.1% Bupivacaine (0.1 ml/kg/hour) both intra- and postoperatively for 24 hours.

Anesthesia was induced with midazolam (0.04 mg/kg), propofol (2 mg/kg) and fentanyl (1mcg/kg) in both groups and the neuromuscular blockage was provided with cisatracurium besilate (0,2 mg/kg). Then, insertion of a double-lumen tracheal tube was performed. After standard patient positioning, localization of the tube was checked with a fiberoptic bronchoscope. Pressure controlled ventilation was used (Primius, Drager, Luebeck, Germany) and invasive arterial pressure, electrocardiography, arterial blood gas analysis, end-tidal carbon dioxide concentration, central venous pressure and urine output were closely monitored in the operating room. Hypothermia was avoided with the help of a warming system and body temperature was kept over 36°C. In TEA group, absolute intraoperative analgesia was warranted with 0,5-2 MAC sevoflurane. In IVA group, remifentanyl infusion (0.1-0.2 mcg/kg/min) was additionally used for this purpose. If arterial pressure exceeds a value of 20% or more of baseline recordings, 1 mcg/kg fentanyl was administered. Every one hour, an additional dose (0.25 mg/kg) of cisatracurium besilate was administered to ensure complete myorelaxation.

The intercostal blockage was applied by the surgical team to the entire population before closing the wound by injecting 4 ml of 0.25% bupivacaine to the region of incision and two intercostal regions above and below the incision site. Once closure was started, morphine sulphate (0,1 mg/kg), tramadol (100 mg), paracetamol (100 mg) and tenoxicam (20 mg) was given intravenously. Anterior 28 Ch and posterior 32 Ch drainage tubes were inserted to the patients to whom lobectomy or bilobectomy was performed. For pneumectomy, only posterior 32 Ch tube was placed. After reversal of neuromuscular blocking agents, patients with adequate spontaneous ventilation and verbal response were transferred to the critical care unit.

Regarding to peri-operative data, procedure time, type of the operation (lobectomy or pneumectomy), duration of tube drainage and presence of operation related complications were recorded.

Visual Analogue Score (VAS) was used to estimate the severity of pain. A score of 0 cm represented "no pain at all" and 10 cm did "intractable pain" so.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists -ASA- Class I to III)
* Scheduled for an elective thoracic surgical procedure with posterolateral thoracotomy

Exclusion Criteria:

* Individuals beyond defined age limits
* Having psychiatric problems
* Having an auditory deficit
* Active drug abuse
* Severe cardiovascular system disorders
* Severe respiratory depression depicted as having less than 50% of the predicted value of forced expiratory volume
* Refusing to give consent
* Contraindication to insertion of an epidural catheter.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 62 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Postoperative FEV1 and FVC alterations | 3 days
  Comparison of preoperative and postoperative FEV1 (liters, %) and FVC.(liters, %)

SECONDARY OUTCOMES:
Postoperative pH alteration | 24 hours
  pH value at 1st and 24th postoperative hours were compared
Postoperative pO2 alteration | 24 hours
  pO2 (mmHg) value at 1st and 24th postoperative hours were compared
Postoperative pCO2 alteration | 24 hours
  pCO2 (mmHg) value at 1st and 24th postoperative hours were compared
Postoperative HCO3 concentration alteration | 24 hours
  Bicarbonate concentration (mEq/dL) at 1st and 24th postoperative hours were compared

IPD SHARING:
Plan to Share IPD: Yes
Can be provided on request
Supporting Information: Study Protocol, ICF, CSR
Time Frame: 1 week
Access Criteria: E-mail

REFERENCES:
- [Result] Erturk E, Aydogdu Kaya F, Kutanis D, Besir A, Akdogan A, Geze S, Tugcugil E. The effectiveness of preemptive thoracic epidural analgesia in thoracic surgery. Biomed Res Int. 2014;2014:673682. doi: 10.1155/2014/673682. Epub 2014 Mar 13. PMID 24745020
- [Result] Helander EM, Webb MP, Bias M, Whang EE, Kaye AD, Urman RD. Use of Regional Anesthesia Techniques: Analysis of Institutional Enhanced Recovery After Surgery Protocols for Colorectal Surgery. J Laparoendosc Adv Surg Tech A. 2017 Sep;27(9):898-902. doi: 10.1089/lap.2017.0339. Epub 2017 Jul 25. PMID 28742434
- [Result] Rawal N. Epidural technique for postoperative pain: gold standard no more? Reg Anesth Pain Med. 2012 May-Jun;37(3):310-7. doi: 10.1097/AAP.0b013e31825735c6. PMID 22531384